CLINICAL TRIAL: NCT07304713
Title: Feasibility and Acceptability of a 12-week Probiotic Intervention to Improve Health Outcomes for People With Multiple Sclerosis: A Single-arm Trial
Brief Title: Probiotic Intervention for People With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Hallam University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ER46295102
Record Dates: First submitted 2025-11-28; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis
Keywords: Feasibility; probiotic; Acceptability; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Mixed-methods
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Probiotic (Experimental): Daily 70ml probiotic
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic — 12-week probiotic intervention (70ml daily)

SUMMARY:
The goal of this single-arm, mixed methods trial is to learn if it is feasible and acceptable to take a probiotic for 12-weeks in people with Multiple Sclerosis. The main question[s] it aims to answer [is/are]:

* Is it feasible and acceptable for people with MS to take a probiotic for 12-weeks?
* Explore impact on health outcomes? Participants will.
* Drink 70ml probiotic drink daily as prescribed for 12-weeks.
* All data collection will be done remotely.
* Before and after 12-weeks participants will complete an online questionnaire (Acceptability, lifestyle behaviour, symptoms, quality of life).
* Provide a stool sample to analyse microbiome changes.
* Take a short online cognitive test.
* Participate in a focus group.

DETAILED DESCRIPTION:
1. Introduction The estimated number of people with MS worldwide has increased to 2.8 million in 2020, with a global prevalence of 35.9 [95% CI: 35.87, 35.95] per 100,000 people. This is estimated to be 30% higher than in 2013 [1].

   Multiple Sclerosis (MS) is a complex and chronic autoimmune disease affecting the central nervous system (CNS). Disease-modifying therapies (DMTs) help manage MS by targeting the immune system to reduce inflammation and nerve damage, thereby lowering relapse rates, MRI lesions, and disability progression. However, their efficacy, safety, and tolerability vary, with significant side effects and limited benefit in progressive MS [2,3]. Long-term self-management of symptoms is therefore a crucial part of treatment.

   The link between the gastrointestinal tract and the brain (i.e., the gut-brain axis) and the increased prevalence of gastrointestinal symptoms across neurological conditions is well known [4,5,6]. The role of the gut microbiome is increasingly being explored in neurological conditions and is of growing interest in MS [7,8,9,10]. In people with MS (PwMS), the gut microbiome is reported to be pathogen-heavy [11], and compositionally and functionally different to healthy controls [12,13]. Many of the diminished bacteria produce short-chain fatty acids (SCFAs), which may drive the chronic inflammation observed in PwMS [12]. These SCFAs are also thought to influence disease onset, re-lapse rates, and overall prognosis [14].

   Probiotics are considered a microbiome-targeted therapy that offers potential for disease management through modulation of the gut microbiome [10]. Current research investigating the potential of probiotics in neurological conditions is still in its infancy, mainly in pre-clinical, animal models or small-scale trials focusing on specific mechanisms or symptoms. The few studies carried out with PwMS demonstrate that certain probiotics may improve symptoms such as poor mental health [15,16]. Recent research has evaluated the impact of probiotics containing Lactiplantibacillus plantarum on MS symptoms, reporting improvements in cognitive impairment, memory and anxiety [15], with research suggesting that approved probiotic supplements should be considered by healthcare professionals to help MS symptom management [10].

   SymproveTM UK is a commercially available probiotic containing Lactiplantibacillus plantarum, in combination with three other bacteria strains, showing promise in other neurodegenerative conditions, such as Parkinsons [18,19]. To date, there is minimal data on the feasibility and acceptability of taking probiotics in PwMS, with initial data suggesting it is tolerated and safe [20].

   The proposed project aimed to assess the feasibility, acceptability, safety and efficacy [21] of running a probiotic (SymproveTM UK) trial with PwMS using a mixed methods approach.
2. Materials and Methods 2.1. Study Design This was a mixed-methods single-arm trial to determine feasibility, acceptability, safety and explore the efficacy of a 12-week probiotic intervention in PwMS. An RCT was not considered necessary at this stage [22], with this approach requiring fewer participants and offering a more cost-effective and ethical approach. This study was approved by the Sheffield Hallam University Research Ethics Committee (ER46295102). An overview of the study design is presented in Figure 1.

2.2. Participants 2.2.1. Sample size Sample sizes of between 12 and 25 per study arm are recommended for feasibility and pilot trial [23,24]. Accounting for an attrition rate of 15-25%, our target sample size was 25-30 participants for this single arm study.

2.2.2. Inclusion and Exclusion Criteria Adults aged 18 years or over, living in the United Kingdom, with a self-reported clinical diagnosis of MS. Exclusion criteria include: a symptom relapse or hospital admission in the prior four weeks; rapidly progressing MS defined as two of more disabling relapses in the last year; immunocompromised and requiring steroids (not including PwMS taking anti-CD20 monoclonal antibodies [Ocrevus or Kesimpta]); type 2 diabetes; cardiovascular disease, kidney disease, chronic gastrointestinal tract health issues; pregnant or lactating; dysphagia; antibiotic use in the prior three months; pro-biotic use in the prior four weeks; use of food supplements which target gut health in the prior four weeks; and if medically advised not to use a probiotic.

2.2.3. Recruitment and Setting Study adverts were disseminated via online MS interest groups and through word of mouth. People who expressed interest in the study were contacted by a researcher to check eligibility. Participant information sheets and consent forms were emailed or posted to potential participants. Informed consent was obtained from all subjects involved in the study using paper or online consent forms. All aspects of the study were conducted remotely. Study documents, assessments and probiotics were posted to participants' preferred address. Prepaid packaging was given to participants to return documents and assessments.

2.3. Intervention Participants were provided with a 12-week supply of original flavour probiotic drink (SymproveTMUK). The probiotic is a water-based, fermented grain beverage containing four strains of live bacteria: Lacticaseibacillus rhamnosus (NCIMB 30174), Enterococcus faecium (NCIMB 30176), Lactobacillus acidophilus (NCIMB 30175), and Lactiplantibacillus plantarum (NCIMB 30173). Providing a total of at least 10 billion Colony Forming Units (CFU) per 70ml serving at the time of manufacture (50% lactobacillus species and 50% enterococcus species).

Participants were required to ingest 70mL of the probiotic drink per day for 84 consecutive days (12-weeks), as soon as possible after waking, on an empty stomach at least 10 minutes before their first meal, late and missed doses were recorded in the adherence diary, with missed doses taken at the end of the 12-weeks. Expected acute side effects of probiotics include increased flatulence, burping, abdominal bloating, abdominal pain or discomfort, constipation and diarrhoea. These side effects are usually mild and transient, typically resolving in the first 2-3 weeks of regular probiotic use. Possible side effect information was conveyed in the participant information sheet and during a telephone call prior to participation.

2.5. Assessments and Outcome Measures 2.5.1 Primary Outcome Measures Recruitment, Retention and Adherence Recruitment, retention and adherence rates were monitored throughout the project. Recruitment was reported as the percentage of eligible participants from those that expressed an interest in the study. Retention was reported as the percentage of participants who completed all aspects of the study. Adherence was monitored with a paper diary, including reasons for missed/late doses.

Safety Participants recorded any potential side effects in a paper diary. In addition, a researcher contacted each participant via telephone or email in the first, second and sixth weeks of the intervention to monitor potential side effects and adverse events in accordance with Good Clinical Practice guidance.

Acceptability The retrospective acceptability of the intervention was assessed after the intervention period using a seven-item questionnaire based on the Theoretical Framework of Acceptability (TFA) [25]. Questionnaire domains include affective attitude, burden, ethicality, intervention coherence, self-efficacy, opportunity cost, and general acceptability. In addition, two online focus groups were conducted to explore acceptability in more detail and obtain qualitative feedback about the study procedures and effects. Focus group interview scripts were guided by the TFA [21,25]. The focus group topic guides were developed by researchers and practitioners working in the sector.

2.5.2. Secondary Outcome Measures Secondary outcome data was collected pre-intervention (week-0) and post-intervention (week-12).

Health-Related Symptom Assessments and Cognitive Function The following outcome measures were assessed at baseline and after the intervention: MS-related quality of life (MSQoL-54) [26], health-related quality of life (EuroQol-5D-3L)[27,28], mental wellbeing (Short Warwick-Edinburgh Mental Wellbeing Scale [SWEMWS])[29], functional ability (Patient Determined Disease Steps[PDDS])[30], gut symptoms (Irritable Bowel Severity Scoring System [IBS-SSS])[31], fatigue (Modified Fatigue Impact Scale [MFIS])[32,33]. Cognitive function was assessed using a self-administered subscale of the Wechsler Adult Intelligence Scale (Fourth UK Edition [WAIS-IV]) [34.35].

Lifestyle Behaviours Participants were asked to maintain their usual lifestyle behaviours during the trial to reduce additional influence on the gut-microbiome. Physical activity and diet were monitored pre- and post-intervention to determine if any significant changes had occurred across the 12-week period that may have impacted on the gut-microbiome. Physical activity levels were assessed using the International Physical Activity Questionnaire Short Form (IPAQ-SF)[36]. Participants also completed a 4-day diet diary (two weekend and two weekdays) before and after the intervention period to determine diet consistency. This was analysed using Nutritics software (Version 6). Nutritics is a cloud-based food data management software platform, offering detailed nutrition analysis

Stool Sample Acceptability The acceptability of taking an at home stool sample was recorded as the number of samples provided and the percentage of samples of sufficient quality for analysis (16s DNA Sequencing). Stool samples were collected before and after the intervention using a commercially available stool sample kit (Biomesight, UK). All samples were collected by participants within seven days of completing the questionnaires, cognitive assessment and 4-day food diary. Stool samples were collected with a swab, then inserted into a collection tube and mixed with a preservative solution for 30 seconds. After discarding the collection swab, the collection tube lid was sealed and shaken vigorously for 10 seconds. The collection tube was then sealed within a specimen bag and posted to the Biomesight laboratory using pre-paid packaging. Samples were preserved with a DNA Shield from Zymo Research and would have remained stable for at least 1-month. All samples were collected and processed within 1-2 weeks, with collection and pro-cessing dates recorded.

Here the investigators reported on the acceptability of this process for PwMS, detailed microbiome analysis is being carried out and will be reported in due course.

2.6. Data Analysis The feasibility, acceptability, safety and preliminary efficacy of the intervention was assessed using a mixed method approach. Theoretical Framework of Acceptability (TFA) questionnaire data are summarised using descriptive statistics. In addition, preliminary hypothesis testing was performed to compare pre-post intervention scores as recommended by Lancaster et al., 2004 [37] for pilot and feasibility research. For para-metric ordinal and continuous data, paired-sample t-tests were used to determine differences between pre- and post-intervention results. Pre-post lifestyle data (physical activity and diet) were assessed as above. Lastly, audio recordings from the focus groups were transcribed verbatim by a third-party transcription company. Deductive thematic analysis [38] was conducted using the seven domains of the TFA as a guide. Three re-searchers then verified and refined themes.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or over.
* Living in the United Kingdom.
* Self-reported clinical diagnosis of MS.

Exclusion Criteria:

* Symptom relapse or hospital admission in the prior four weeks.
* Rapidly progressing MS defined as two of more disabling relapses in the last year.
* Immunocompromised and requiring steroids (not including PwMS taking anti-CD20 monoclonal antibodies [Ocrevus or Kesimpta]).
* Type 2 diabetes, Cardiovascular disease, kidney disease, chronic gastrointestinal tract health issues.
* Pregnant or lactating.
* Dysphagia.
* Antibiotic use in the prior three months.
* Pro-biotic use in the prior four weeks.
* Use of food supplements which target gut health in the prior four weeks.
* Medically advised not to use a probiotic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2023-11-24 (Actual); Study Completion 2023-11-24 (Actual)

PRIMARY OUTCOMES:
Recruitment | 8-weeks
  Percentage of eligible participants recruited from those who had expressed interest.
Retention | 23-weeks
  Percentage of participants who completed all aspects of the study.
Adherence | 12-weeks
  Described as the percentage of doses taken. This was recorded with a paper diary and contained information on reason for missed/late doses.
Safety/Side effects | 12-weeks
  Participants recorded all potential side effects in a diary, as well as being asked by the researcher at 1,2 and 6 weeks.
Acceptability | 0-weeks (baseline) and 12-week (Follow-up)
  Acceptability was measured using the 7 domains of the Sehkon acceptability framework, both via self-report questionnaire on the Qualtrics platform and during online qualitative focus groups.

SECONDARY OUTCOMES:
Overall Quality of life of participants | Baseline (0-weeks) and Follow-up (12-week)
  Multiple Sclerosis related quality of life (MSQoL-54). Assessed by self-report questionnaire on the Qualtrics platform. The scoring method uses weighted calculations based on the patient's answers. The questionnaire gathers data through Likert scales, multiple-choice, yes/no, and rating scale questions. Scores for each domain are converted to a 0-100 scale. Scoring procedures generate two primary composite scores: the Physical Health Composite and the Mental Health Composite. A higher score indicates a better health-related quality of life (HRQOL). Conversely, lower scores indicate poorer HRQOL.
Health-related quality of life | Baseline (0-weeks) and Follow-up (12-weeks)
  Health Related Quality of Life (EuroQol-5D 3L). Assessed by self-report questionnaire on the Qualtrics platform. The EQ-5D-3L consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state', 0 to 100. The VAS can be used as a quantitative measure of health.
Participant mental wellbeing | Baseline (0-weeks) and Follow-up (12 weeks)
  Short Warwick-Edinburgh mental wellbeing scale (WEMWBS). Assessed by self-report questionnaire on the Qualtrics platform. The WEMWBS is scored by summing the scores for each of the 14 items, which are scored from 1 to 5. Total scores are summed and range from 14 to 70. Higher scores are associated with higher levels of mental wellbeing.
Participant functional ability | Baseline (0-weeks) and Follow-up (12-weeks)
  Patient Determined Disease Steps (PDDS). Assessed by self-report questionnaire on the Qualtrics platform. PDDS scores correlate with mobility, dexterity, and fatigue in older adults with MS. Higher PDDS scores are associated with lower grey matter volume in key brain regions. The PDDS is a valid self-report measure of disability in ambulatory older adults with MS.
Participant Gut Symptoms | Baseline (0-weeks) and Follow-up (12-weeks)
  Irritable Bowel Severity Scoring System (IBS-SSS). The IBS-SSS questionnaire evaluates five key areas: Pain Severity, Pain Frequency, Bloating, Bowel Dysfunction, Quality of Life. Scores are rated on a scale from 0 to 100, with lowers scores indicating better health.
Participant fatigue | Baseline (0-weeks) and Follow-up (12-weeks).
  Modified Fatigue Impact Scale (MFIS). The MFIS is a self-report questionnaire and was delivered online using Qualtrics designed to measure the impact of fatigue on various aspects of life in individuals with MS. The MFIS consists of 21 items divided into three subscales: Physical, Cognitive and Psychosocial. Respondents rate each item on a scale from 0 (no problem) to 4 (extreme problem), with higher scores indicating a greater impact of fatigue. The total score ranges from 0 to 84.
Cognitive function (processing speed) | Baseline (0-weeks) and Follow-up (12-weeks)
  Subscale of the Wechsler Adult Intelligence Scale (WAIS-IV). Processing Speed Index was measured at home following instructions and using a paper based form. This index reflects an individual's ability to process simple or routine visual information quickly and efficiently and is scored based on the number completed in a set time. The higher the score the better.

OTHER OUTCOMES:
Physical Activity | Baseline (0-weeks) and Follow-up (12-weeks)
  International Physical Activity Questionnaire - Short Form (IPAQ-SF). A self-report questionnaire was used, delivered on the Qualtrics platform. The questionnaire is structured to provide separate scores on the amount of time spent walking; doing moderate-intensity; and vigorous-intensity activity in a week, with a combined total score used to describe overall level of physical activity. A higher score indicates greater levels of physical activity.
Diet Diary | Baseline (0-weeks) and Follow-up (12-weeks)
  Four day diet diary, consisting of two weekdays and two weekend days. Results were analysed using Nutritics software to determine if there was any significant differences in nutritional content and overall calorie consumption.
Stool sample acceptability | Baseline (0-weeks) and Follow-up (12-weeks)
  Acceptability of taking samples, measured as percentage of quality samples obtained.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Hallam University, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No